CLINICAL TRIAL: NCT01447225
Title: A Phase 1, Pharmacologic and Pharmacodynamic Study of MM-121 in Combination With Multiple Anticancer Therapies in Patients With Advanced Solid Tumors
Brief Title: Safety Study of MM-121 in Combination With Multiple Anticancer Therapies in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-121-06-01-06 (TCD11694)
Record Dates: First submitted 2011-10-03; First posted 2011-10-06 (Estimated); Results first posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Solid Tumors
Keywords: Advanced-stage; Solid Tumors; MM-121; Carboplatin; Pemetrexed; Gemcitabine; Cabazitaxel; ErbB3; Phase I; Cancer
MeSH Terms: conditions — Neoplasms | interventions — seribantumab; Carboplatin; Pemetrexed; cabazitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MM-121 plus Gemcitabine (Experimental): escalating doses of MM-121 and gemcitabine on Day 1 and Day 8 of every 3 week cycle
  Interventions: Drug: MM-121; Drug: Gemcitabine
- MM-121 plus Carboplatin (Experimental): carboplatin at AUC 6 with escalating doses of MM-121 on Day 1 of every 3 week cycle
  Interventions: Drug: MM-121; Drug: Carboplatin
- MM-121 plus Pemetrexed (Experimental): pemetrexed at 500 mg/m2 with escalating doses of MM-121 on Day 1 of every 3 week cycle
  Interventions: Drug: MM-121; Drug: Pemetrexed
- MM-121 plus Cabazitaxel (Experimental): escalating doses of MM-121 and cabazitaxel on Day 1 of every 3 week cycle
  Interventions: Drug: MM-121; Drug: Cabazitaxel

INTERVENTIONS:
Drug: MM-121 — MM-121 administered at 20 mg/kg IV loading dose followed by12mg/kg/week IV or 40 mg/kg IV loading dose followed by 20mg/kg/week IV
  Other Names: Seribantumab, SAR256212
Drug: Carboplatin — administered at AUC 6
  Arms: MM-121 plus Carboplatin
Drug: Pemetrexed — administered IV at 500 mg/m2
  Other Names: ALIMTA
  Arms: MM-121 plus Pemetrexed
Drug: Cabazitaxel — administered IV at 20 mg/m2 or 25 mg/m2
  Other Names: Jevtana
  Arms: MM-121 plus Cabazitaxel
Drug: Gemcitabine — administered IV at 1000 mg/m2 or 1250 mg/m2
  Other Names: Gemzar
  Arms: MM-121 plus Gemcitabine

SUMMARY:
To evaluate the safety and tolerability of escalating doses of MM-121 + certain anticancer therapies

DETAILED DESCRIPTION:
This study was a Phase 1 and pharmacologic dose-escalation trial of MM-121 in combination with certain anticancer therapies. The dose-escalation portion of the study employed a 3 + 3 design to assess the safety, tolerability, and pharmacokinetics of MM-121 administered weekly in combination with certain anticancer therapies in patients with advanced/recurrent cancer. Doses of MM-121 and/or the anticancer therapy were escalated until either the MTD is identified or the combination was shown to be tolerable at the highest planned doses.

ELIGIBILITY:
Inclusion Criteria:

* Advanced-stage solid tumors
* ≥ 18 years of age
* Adequate liver and kidney function

Exclusion Criteria:

* Any other active malignancy
* No known HIV, Hepatitis C or B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Moyo, MD, Study Director — Merrimack Pharmaceuticals
Locations (5):
- United States (4):
  - Lafayette, Indiana
  - Buffalo, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
- Villejuif, France

RESULTS

PARTICIPANT FLOW:
Groups:
- MM-121 Plus Gemcitabine: Cohort 1: MM-121 20 mg/kg one-time loading dose on Cycle 1, Week 1 followed 12 mg/kg IV maintenance doses weekly for 3-week cycles
  gemcitabine 1000 mg/m2 IV on Days 1 and 8 of each 3-week cycle
- MM-121 Plus Gemcitabine: Cohort 2: MM-121 40 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 20 mg/kg IV maintenance doses weekly for each 3-week cycle
  Gemcitabine: 1000 mg/m2 IV on Day 1 And Day 8 of each 3-week cycle
- MM-121 Plus Carboplatin: Cohort 1: MM-121: 20 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 12 mg/kg IV maintenance doses weekly for each 3-week cycle
  Carboplatin at AUC 6 Day 1 of every 3 week cycle
- MM-121 Plus Carboplatin: Cohort 2: MM-121: 20 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 12 mg/kg IV maintenance doses weekly for each 3-week cycle
  Carboplatin at AUC 5 Day 1 of every 3 week cycle
- MM-121 Plus Carboplatin: Cohort 3: MM-121: 40 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 20 mg/kg IV maintenance doses weekly for each 3-week cycle
  Carboplatin at AUC 5 Day 1 of every 3 week cycle
- MM-121 Plus Pemetrexed: Cohort 1: MM-121: 20 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 12 mg/kg IV maintenance dose weekly for every 3-week cycle
  Pemetrexed at 500 mg/m2 IV on Day 1 of every 3 week cycle
- MM-121 Plus Pemetrexed: Cohort 2: MM-121: 40 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 20 mg/kg IV maintenance dose weekly for every 3-week cycle
  Pemetrexed at 500 mg/m2 IV on Day 1 of every 3 week cycle
- MM-121 Plus Cabazitaxel: Cohort 1: MM-121: 20 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 12mg/kg IV maintenance doses weekly for each 3-week cycle
  Cabazitaxel: 20 mg/m2 IV on Day 1 of each 3-week cycle
- MM-121 Plus Cabazitaxel: Cohort 2: MM-121: 40 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 20 mg/kg maintenance doses weekly for each 3-week cycle
  Cabazitaxel: 20 mg/m2 IV on Day 1 of each 3-week cycle
- MM-121 Plus Cabazitaxel: Cohort 3: MM-121: 40 mg/kg IV one-time loading dose on Cycle 1, Week 1 followed by 20 mg/kg maintenance doses weekly for each 3-week cycle
  Cabazitaxel: 25 mg/m2 IV on Day 1 of each 3-week cycle
Period: Overall Study
Arm/Group | MM-121 Plus Gemcitabine: Cohort 1 | MM-121 Plus Gemcitabine: Cohort 2 | MM-121 Plus Carboplatin: Cohort 1 | MM-121 Plus Carboplatin: Cohort 2 | MM-121 Plus Carboplatin: Cohort 3 | MM-121 Plus Pemetrexed: Cohort 1 | MM-121 Plus Pemetrexed: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 1 | MM-121 Plus Cabazitaxel: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 3
Started | 3 | 8 | 5 | 3 | 3 | 3 | 7 | 4 | 3 | 4
Completed | 3 | 8 | 5 | 3 | 3 | 3 | 7 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MM-121 Plus Gemcitabine | MM-121 Plus Carboplatin | MM-121 Plus Pemetrexed | MM-121 Plus Cabazitaxel | Total
Number analyzed (Participants) | 11 | 11 | 10 | 11 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (7.79) | 62.7 (9.18) | 60.0 (12.29) | 64.1 (6.66) | 61.28 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 7 | 2 | 22
  Male | 3 | 6 | 3 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 10 | 11 | 10 | 11 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 11 | 9 | 11 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 7 | 8 | 34
  France | 3 | 0 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety and Tolerability of Escalating Doses of the MM-121 Anticancer Therapies
Description: Safety and tolerability data presented in detail in the adverse events and serious adverse events section of the results posting
Time Frame: From date of first dose to 30 days after termination, the longest 88.1 weeks
Measure: Number; unit: participants reporting adverse events
Arm/Group | MM-121 Plus Gemcitabine: Cohort 1 | MM-121 Plus Gemcitabine: Cohort 2 | MM-121 Plus Carboplatin: Cohort 1 | MM-121 Plus Carboplatin: Cohort 2 | MM-121 Plus Carboplatin: Cohort 3 | MM-121 Plus Pemetrexed: Cohort 1 | MM-121 Plus Pemetrexed: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 1 | MM-121 Plus Cabazitaxel: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 3
Number analyzed (Participants) | 3 | 8 | 5 | 3 | 3 | 3 | 7 | 4 | 3 | 4
participants reporting adverse events | 3 | 8 | 5 | 3 | 3 | 3 | 7 | 4 | 3 | 4

2. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of MM-121 in Combination With Anticancer Therapies: MM-121 Doses
Description: Using a 3+3 dose escalation model, the maximum tolerated dose of each therapy combination was determined by assessing dose-limiting toxicities in each cohort. If 3 patients were treated and passed the observation window, escalation to the next cohort was initiated. If a DLT was reported, 3-4 additional patients were enrolled and observed. If a DLT was observed in expanded cohort, this dose was considered to be the maximum tolerated dose. The maximum tolerated dose was defined at the cohort in which two dose-limiting toxicities were observed, or as the highest target dose tested in the absence of DLTs. The determined MTD was considered the Recommended Phase 2 Dose.
  Dose Levels (3 week cycles) MM-121 doses tested: 20 mg/kg IV one-time loading dose then 12 mg/kg IV QW (20/12 mg/kg); 40/20 mg/kg Gemcitabine doses tested: 1000 mg/m2 Day 1 and 8 Pemetrexed doses tested: 500 mg/m2 Day 1 Carboplatin doses tested: 5 or 6 AUC Day 1 Cabazitaxel doses tested: 20 or 25 mg/m2 Day 1 of 3
Time Frame: From date of first dose to 30 days after termination, the longest 88.1 weeks
Population: Note: data provided below is for MM-121 doses only for the combination. Combination therapy MTDs are provided in separate endpoint measures.
Measure: Number; unit: mg/kg
Arm/Group | MM-121 Plus Gemcitabine | MM-121 Plus Carboplatin | MM-121 Plus Pemetrexed | MM-121 Plus Cabazitaxel
Number analyzed (Participants) | 11 | 11 | 10 | 11
mg/kg
  one-time loading dose | 40 | 40 | 40 | 40
  maintenance dose | 20 | 20 | 20 | 20

3. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of MM-121 in Combination With Anticancer Therapies: Gemcitabine
Description: Using a 3+3 dose escalation model, the maximum tolerated dose of each therapy combination was determined by assessing dose-limiting toxicities in each cohort. If 3 patients were treated and passed the observation window, escalation to the next cohort was initiated. If a DLT was reported, 3-4 additional patients were enrolled and observed. If a DLT was observed in expanded cohort, this dose was considered to be the maximum tolerated dose. The maximum tolerated dose was defined at the cohort in which two dose-limiting toxicities were observed, or as the highest target dose tested in the absence of DLTs. The determined MTD was considered the Recommended Phase 2 Dose.
  Dose Levels (3 week cycles) MM-121 doses tested: 20 mg/kg IV one-time loading dose then 12 mg/kg IV QW (20/12 mg/kg); 40/20 mg/kg Gemcitabine doses tested: 1000 mg/m2 Day 1 and 8
Time Frame: From date of first dose to 30 days after termination, the longest 88.1 weeks
Population: NOTE: Maximum tolerated dose is for the combination of gemcitabine and MM-121. MTD of MM-121 is provided in separate endpoint.
Measure: Number; unit: mg/m2
Arm/Group | MM-121 + Gemcitabine
Number analyzed (Participants) | 11
mg/m2 | 1000

4. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of MM-121 in Combination With Anticancer Therapies: Carboplatin
Description: Maximum Tolerated Dose reported in Target AUC, as calculated by the Calvert Formula
  Using a 3+3 dose escalation model, the maximum tolerated dose of each therapy combination was determined by assessing dose-limiting toxicities in each cohort. If 3 patients were treated and passed the observation window, escalation to the next cohort was initiated. If a DLT was reported, 3-4 additional patients were enrolled and observed. If a DLT was observed in expanded cohort, this dose was considered to be the maximum tolerated dose. The maximum tolerated dose was defined at the cohort in which two dose-limiting toxicities were observed, or as the highest target dose tested in the absence of DLTs. The determined MTD was considered the Recommended Phase 2 Dose.
  Dose Levels (3 week cycles) MM-121 doses tested: 20 mg/kg IV one-time loading dose then 12 mg/kg IV QW (20/12 mg/kg); 40/20 mg/kg Carboplatin doses tested: 5 or 6 AUC Day 1
Time Frame: From date of first dose to 30 days after termination, the longest 88.1 weeks
Measure: Number; unit: target AUC (mg*min/mL)
Groups:
- MM-121 + Carboplatin: MTD of the MM-121 + Carboplatin combination NOTE: MTD of MM-121 for this combination provided in separate endpoint
Arm/Group | MM-121 + Carboplatin
Number analyzed (Participants) | 11
target AUC (mg*min/mL) | 5

5. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of MM-121 in Combination With Anticancer Therapies: Pemetrexed
Description: Using a 3+3 dose escalation model, the maximum tolerated dose of each therapy combination was determined by assessing dose-limiting toxicities in each cohort. If 3 patients were treated and passed the observation window, escalation to the next cohort was initiated. If a DLT was reported, 3-4 additional patients were enrolled and observed. If a DLT was observed in expanded cohort, this dose was considered to be the maximum tolerated dose. The maximum tolerated dose was defined at the cohort in which two dose-limiting toxicities were observed, or as the highest target dose tested in the absence of DLTs. The determined MTD was considered the Recommended Phase 2 Dose.
  Dose Levels (3 week cycles) MM-121 doses tested: 20 mg/kg IV one-time loading dose then 12 mg/kg IV QW (20/12 mg/kg); 40/20 mg/kg Pemetrexed doses tested: 500 mg/m2 Day 1
Time Frame: From date of first dose to 30 days after termination, the longest 88.1 weeks
Measure: Number; unit: mg/m2
Groups:
- MM-121 + Pemetrexed: MTD of combination of MM-121 + Pemetrexed - NOTE: MTD of MM-121 for this combination provided in separate endpoint
Arm/Group | MM-121 + Pemetrexed
Number analyzed (Participants) | 10
mg/m2 | 500

6. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of MM-121 in Combination With Anticancer Therapies: Cabazitaxel
Description: Using a 3+3 dose escalation model, the maximum tolerated dose of each therapy combination was determined by assessing dose-limiting toxicities in each cohort. If 3 patients were treated and passed the observation window, escalation to the next cohort was initiated. If a DLT was reported, 3-4 additional patients were enrolled and observed. If a DLT was observed in expanded cohort, this dose was considered to be the maximum tolerated dose. The maximum tolerated dose was defined at the cohort in which two dose-limiting toxicities were observed, or as the highest target dose tested in the absence of DLTs. The determined MTD was considered the Recommended Phase 2 Dose.
  Dose Levels (3 week cycles) MM-121 doses tested: 20 mg/kg IV one-time loading dose then 12 mg/kg IV QW (20/12 mg/kg); 40/20 mg/kg Cabazitaxel doses tested: 20 or 25 mg/m2 Day 1 of 3
Time Frame: From date of first dose to 30 days after termination, the longest 88.1 weeks
Measure: Number; unit: mg/m2
Groups:
- MM-121 + Cabazitaxel: MTD of MM-121 + Cabazitaxel combination - NOTE: MTD of MM-121 for this combination provided in separate endpoint
Arm/Group | MM-121 + Cabazitaxel
Number analyzed (Participants) | 11
mg/m2 | 25

7. Primary Outcome: To Characterize Dose-limiting Toxicities (DLTs) Associated With the Combination of MM-121 With Anticancer Therapies
Description: To establish the safety of escalating doses of MM-121 administered in combination with multiple anti-cancer therapies in order to determine the recommended phase 2 dose. Dose-escalation conducted using standard 3+3 model to determine maximum tolerated dose. Reports of Dose-Limiting Toxicities (DLTs) were assessed to determine the MTD to be used for the expansion cohort. DLTs were not measured in the Expansion Cohort.
Time Frame: From date of first dose to 30 days after termination, the longest 88.1 weeks
Measure: Number; unit: participants reporting DLTs
Arm/Group | MM-121 Plus Gemcitabine: Cohort 1 | MM-121 Plus Gemcitabine: Cohort 2 | MM-121 Plus Carboplatin: Cohort 1 | MM-121 Plus Carboplatin: Cohort 2 | MM-121 Plus Carboplatin: Cohort 3 | MM-121 Plus Pemetrexed: Cohort 1 | MM-121 Plus Pemetrexed: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 1 | MM-121 Plus Cabazitaxel: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 3
Number analyzed (Participants) | 3 | 8 | 5 | 3 | 3 | 3 | 7 | 4 | 3 | 3
participants reporting DLTs | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

8. Secondary Outcome: Objective Response Rate
Description: To determine the number of patients reporting an objective response using RECIST v 1.1 where a Partial Response (PR) is defined as >20% decrease in tumor burden from baseline and a Complete Response (CR) is defined as complete disappearance from tumor burden from baseline. Objective Response is presented as the total # patients with PR or CR.
Time Frame: patients were assessed for response during their time on study, the longest of which was 88.1 weeks
Measure: Number; unit: participants with objective response
Arm/Group | MM-121 Plus Gemcitabine: Cohort 1 | MM-121 Plus Gemcitabine: Cohort 2 | MM-121 Plus Carboplatin: Cohort 1 | MM-121 Plus Carboplatin: Cohort 2 | MM-121 Plus Carboplatin: Cohort 3 | MM-121 Plus Pemetrexed: Cohort 1 | MM-121 Plus Pemetrexed: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 1 | MM-121 Plus Cabazitaxel: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 3
Number analyzed (Participants) | 3 | 8 | 5 | 3 | 3 | 3 | 7 | 4 | 3 | 4
participants with objective response | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1

9. Secondary Outcome: Pharmacokinetics
Description: Pharmacokinetic (PK) evaluation was performed on plasma samples obtained weekly for the first cycle of the study and then on day 1 of each additional cycle to assess pre-treatment trough concentrations of MM-121. Non-compartmental analysis (NCA) was performed to calculate standard PK parameters, including the maximum observed concentration (Cmax). Serum levels of MM-121 were measured at a central lab using an enzyme-linked immunosorbent assay (ELISA). Data is presented per dose level of MM-121 (12 mg/kg, 20 mg/kg, or 40/20 mg/kg).
Time Frame: Collections taken at Cycle 1, Week 1 for all patients at start of the infusion (pretreatment), at the end of the infusion, and at 2, 4, 24 and 48 hours after the start of the MM-121 infusion
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- MM-121 + Gemcitabine: 20/12 mg/kg: MM-121 20 mg/kg loading dose followed by 12 mg/kg weekly maintenance dose plus gemcitabine 1000mg/m² or 1250mg/m²
- MM-121 + Carboplatin: 20/12 mg/kg: MM-121 20 mg/kg loading dose followed by 12 mg/kg weekly maintenance dose Plus carboplatin AUC 6
- MM-121 + Pemetrexed: 20/12 mg/kg: MM-121 20 mg/kg loading dose followed by 12 mg/kg weekly maintenance dose Plus pemetrexed 500 mg/m²
- MM-121 + Cisplatin: 20/12 mg/kg: MM-121 20 mg/kg loading dose followed by 12 mg/kg weekly maintenance dose Plus Cisplatin 20 mg/m2 or 25 mg/m2
- MM-121 + Gemcitabine: 40/20 mg/kg: MM-121 40 mg/kg loading dose followed by 20 mg/kg weekly maintenance dose plus gemcitabine 1000mg/m² or 1250mg/m²
- MM-121 + Carboplatin: 40/20 mg/kg: MM-121 40 mg/kg loading dose followed by 20 mg/kg weekly maintenance dose Plus carboplatin AUC 6
- MM-121 + Pemetrexed: 40/20 mg/kg: MM-121 40 mg/kg loading dose followed by 20 mg/kg weekly maintenance dose Plus pemetrexed 500 mg/m²
- MM-121 + Cisplatin: 40/20 mg/kg: MM-121 40 mg/kg loading dose followed by 20 mg/kg weekly maintenance dose Plus Cisplatin 25 mg/m2
Arm/Group | MM-121 + Gemcitabine: 20/12 mg/kg | MM-121 + Carboplatin: 20/12 mg/kg | MM-121 + Pemetrexed: 20/12 mg/kg | MM-121 + Cisplatin: 20/12 mg/kg | MM-121 + Gemcitabine: 40/20 mg/kg | MM-121 + Carboplatin: 40/20 mg/kg | MM-121 + Pemetrexed: 40/20 mg/kg | MM-121 + Cisplatin: 40/20 mg/kg
Number analyzed (Participants) | 3 | 8 | 3 | 4 | 8 | 3 | 7 | 7
ug/mL | 560 (45.2) | 554.8 (30.2) | 900.7 (37.6) | 677.1 (24.0) | 1033.4 (24.2) | 1107.2 (18.3) | 1100.8 (18.0) | 1087.9 (18.2)

10. Secondary Outcome: Pharmacokinetics (AUClast)
Description: Pharmacokinetic (PK) evaluation was performed on plasma samples obtained weekly for the first cycle of the study and then on day 1 of each additional cycle to assess pre-treatment trough concentrations of MM-121. Non-compartmental analysis (NCA) was performed to calculate standard PK parameters, including the AUClast. Serum levels of MM-121 were measured at a central lab using an enzyme-linked immunosorbent assay (ELISA). Data is presented per dose level of MM-121 (12 mg/kg, 20 mg/kg, or 40/20 mg/kg) and per study part (Part 1 or Part 2).
Time Frame: Collections taken at Cycle 1, Week 1 for all patients at the start of the infusion (pretreatment), at the end of the infusion, and at 2, 4, 24 and 48 hours after the start of the MM-121 infusion
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr* ug/mL
Arm/Group | MM-121 + Gemcitabine: 20/12 mg/kg | MM-121 + Carboplatin: 20/12 mg/kg | MM-121 + Pemetrexed: 20/12 mg/kg | MM-121 + Cisplatin: 20/12 mg/kg | MM-121 + Gemcitabine: 40/20 mg/kg | MM-121 + Carboplatin: 40/20 mg/kg | MM-121 + Pemetrexed: 40/20 mg/kg | MM-121 + Cisplatin: 40/20 mg/kg
Number analyzed (Participants) | 3 | 8 | 3 | 4 | 8 | 3 | 7 | 7
hr* ug/mL | 39666.4 (41.0) | 49749.6 (41.3) | 59984.1 (36.9) | 51995.1 (71.1) | 72132.1 (41.9) | 100309.9 (34.2) | 92732.9 (31.1) | 98142.6 (18.0)

11. Secondary Outcome: Immunogenicity
Description: Samples were collected to determine the presence of an immunologic reaction to MM-121 (i.e. human anti-human antibodies).
Time Frame: Samples were collected for all patients pre-dose on all cycles for duration of treatment, the longest of which was 88.1 weeks, and a collection was made post-infusion in any case of infusion reaction
Measure: Number
Arm/Group | MM-121 Plus Gemcitabine: Cohort 1 | MM-121 Plus Gemcitabine: Cohort 2 | MM-121 Plus Carboplatin: Cohort 1 | MM-121 Plus Carboplatin: Cohort 2 | MM-121 Plus Carboplatin: Cohort 3 | MM-121 Plus Pemetrexed: Cohort 1 | MM-121 Plus Pemetrexed: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 1 | MM-121 Plus Cabazitaxel: Cohort 2 | MM-121 Plus Cabazitaxel: Cohort 3
Number analyzed (Participants) | 3 | 8 | 5 | 3 | 3 | 3 | 7 | 4 | 3 | 4
Value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value | NA — The very small number of patients in each cohort and the very low levels of positivity resulted in a non-reportable value

ADVERSE EVENTS:
Time Frame: AEs were collected from a patient's first dose until 30 days after treatment termination. SAEs were collected from time of informed consent until 30 days after termination. If related, events could be reported at any time after termination.
Description: All related AEs ongoing at the time of treatment discontinuation were followed until resolution. Investigators were to report any AEs/SAEs assumed to be related any time, even if occurring more than 30 days after last dose. Though different for each patient, on average, patients could be followed for related AEs/SAEs for ~1 year after termination
Arm/Group | MM-121 Plus Gemcitabine | MM-121 Plus Carboplatin | MM-121 Plus Pemetrexed | MM-121 Plus Cabazitaxel
Serious Adverse Events (participants affected / at risk) | 9/11 | 7/11 | 3/10 | 2/11
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11 | 10/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MM-121 Plus Gemcitabine (N=11) | MM-121 Plus Carboplatin (N=11) | MM-121 Plus Pemetrexed (N=10) | MM-121 Plus Cabazitaxel (N=11)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 — Any Relationship
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 — Any Relationship
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 — Any Relationship
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — Any Relationship
CELLULITIS (Infections and infestations) | 1 | 0 | 1 | 1 — Any Relationship
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 — Any Relationship
ABSCESS LIMB (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
GROIN ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 — Any Relationship
ERYSIPELAS (Infections and infestations) | 0 | 0 | 1 | 0 — Any Relationship
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Any Relationship
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 | 0 | 0 | 0 — Any Relationship
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Any Relationship
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 — Any Relationship
ATAXIA (Nervous system disorders) | 1 | 0 | 0 | 0 — Any Relationship
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0 | 0 — Any Relationship
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1 | 0 | 0 — Any Relationship
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0 — Any Relationship
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 — Any Relationship
EMBOLISM (Vascular disorders) | 0 | 1 | 0 | 0 — Any Relationship
DISEASE PROGRESSION (General disorders) | 0 | 1 | 0 | 0 — Any Relationship
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 1 | 0 — Any Relationship
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1 | 0 — Any Relationship
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 1 — Any Relationship
CENTRAL VENOUS CATHETER REMOVAL (Surgical and medical procedures) | 0 | 0 | 1 | 0 — Any Relationship
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MM-121 Plus Gemcitabine (N=11) | MM-121 Plus Carboplatin (N=11) | MM-121 Plus Pemetrexed (N=10) | MM-121 Plus Cabazitaxel (N=11)
NAUSEA (Gastrointestinal disorders) | 7 | 8 | 4 | 7 — Any Relationship
DIARRHOEA (Gastrointestinal disorders) | 6 | 9 | 7 | 11 — Any Relationship
VOMITING (Gastrointestinal disorders) | 6 | 6 | 2 | 3 — Any Relationship
CONSTIPATION (Gastrointestinal disorders) | 4 | 2 | 2 | 2 — Any Relationship
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 1 | 1 | 1 — Any Relationship
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2 | 2 | 1 — Any Relationship
STOMATITIS (Gastrointestinal disorders) | 3 | 1 | 2 | 4 — Any Relationship
ABDOMINAL RIGIDITY (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 1 | 0 — Any Relationship
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 1 | 0 | 0 — Any Relationship
HIATUS HERNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
FLATULENCE (Gastrointestinal disorders) | 0 | 2 | 0 | 1 — Any Relationship
ASCITES (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
BREATH ODOR (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 3 — Any Relationship
ODYNOPHAGIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
PAINFUL DEFAECATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 1 — Any Relationship
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 2 — Any Relationship
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 2 — Any Relationship
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 2 — Any Relationship
CHAPPED LIPS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Any Relationship
URINARY TRACT INFECTION (Infections and infestations) | 4 | 3 | 1 | 1 — Any Relationship
CELLULITIS (Infections and infestations) | 2 | 0 | 1 | 2 — Any Relationship
ORAL FUNGAL INFECTION (Infections and infestations) | 2 | 0 | 1 | 0 — Any Relationship
PNEUMONIA (Infections and infestations) | 2 | 0 | 0 | 2 — Any Relationship
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2 | 0 | 4 — Any Relationship
EAR INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 — Any Relationship
FUNGAL SKIN INFECTION (Infections and infestations) | 1 | 0 | 1 | 0 — Any Relationship
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 — Any Relationship
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 0 | 0 — Any Relationship
RASH PUSTULAR (Infections and infestations) | 1 | 0 | 0 | 0 — Any Relationship
RHINITIS (Infections and infestations) | 1 | 0 | 1 | 0 — Any Relationship
SINUSITIS (Infections and infestations) | 1 | 1 | 0 | 0 — Any Relationship
TINEA PEDIS (Infections and infestations) | 1 | 0 | 0 | 0 — Any Relationship
ABSCESS LIMB (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
BRONCHITIS (Infections and infestations) | 0 | 1 | 0 | 1 — Any Relationship
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 1 — Any Relationship
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
GROIN ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 — Any Relationship
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 — Any Relationship
ERYSIPELAS (Infections and infestations) | 0 | 0 | 1 | 0 — Any Relationship
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 — Any Relationship
PARONYCHIA (Infections and infestations) | 0 | 0 | 0 | 3 — Any Relationship
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 1 — Any Relationship
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 1 — Any Relationship
URETERITIS (Infections and infestations) | 0 | 0 | 0 | 1 — Any Relationship
FATIGUE (General disorders) | 5 | 6 | 7 | 5 — Any Relationship
OEDEMA PERIPHERAL (General disorders) | 4 | 2 | 4 | 3 — Any Relationship
PYREXIA (General disorders) | 4 | 1 | 2 | 1 — Any Relationship
MUCOSAL INFLAMMATION (General disorders) | 3 | 1 | 1 | 4 — Any Relationship
ASTHENIA (General disorders) | 2 | 0 | 3 | 5 — Any Relationship
CHILLS (General disorders) | 1 | 0 | 2 | 2 — Any Relationship
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0 | 3 — Any Relationship
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 1 | 0 | 0 — Any Relationship
OEDEMA (General disorders) | 1 | 0 | 0 | 0 — Any Relationship
PAIN (General disorders) | 1 | 0 | 0 | 0 — Any Relationship
SUPRAPUBIC PAIN (General disorders) | 1 | 0 | 0 | 0 — Any Relationship
XEROSIS (General disorders) | 1 | 0 | 0 | 1 — Any Relationship
CATHETER SITE RASH (General disorders) | 0 | 1 | 0 | 0 — Any Relationship
DISEASE PROGRESSION (General disorders) | 0 | 1 | 0 | 0 — Any Relationship
CHEST PAIN (General disorders) | 0 | 0 | 1 | 1 — Any Relationship
INJECTION SITE HAEMORRHAGE (General disorders) | 0 | 0 | 1 | 0 — Any Relationship
EARLY SATIETY (General disorders) | 0 | 0 | 0 | 1 — Any Relationship
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 1 — Any Relationship
INJECTION SITE PAIN (General disorders) | 0 | 0 | 0 | 1 — Any Relationship
ANAEMIA (Blood and lymphatic system disorders) | 7 | 5 | 4 | 6 — Any Relationship
NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 0 | 3 | 4 — Any Relationship
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 5 | 1 | 4 — Any Relationship
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 — Any Relationship
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 | 0 | 1 | 3 — Any Relationship
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 — Any Relationship
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 — Any Relationship
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 — Any Relationship
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — Any Relationship
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — Any Relationship
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 | 3 | 3 | 4 — Any Relationship
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 2 | 3 | 6 — Any Relationship
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 4 | 2 | 1 | 7 — Any Relationship
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 1 | 1 | 4 — Any Relationship
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 — Any Relationship
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 | 3 | 2 | 3 — Any Relationship
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 — Any Relationship
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2 — Any Relationship
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 — Any Relationship
GOUT (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Any Relationship
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Any Relationship
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 — Any Relationship
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 — Any Relationship
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 — Any Relationship
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 — Any Relationship
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 — Any Relationship
POLYDIPSIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 — Any Relationship
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 1 — Any Relationship
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 4 — Any Relationship
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 2 — Any Relationship
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 — Any Relationship
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 — Any Relationship
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 — Any Relationship
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Any Relationship
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 — Any Relationship
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Any Relationship
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — Any Relationship
DYSPNOAE EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Any Relationship
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Any Relationship
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Any Relationship
NOCTURNAL DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Any Relationship
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Any Relationship
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 — Any Relationship
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 2 — Any Relationship
RASH (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 3 — Any Relationship
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Any Relationship
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 — Any Relationship
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 — Any Relationship
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 — Any Relationship
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 — Any Relationship
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 — Any Relationship
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Any Relationship
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 — Any Relationship
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Any Relationship
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 — Any Relationship
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Any Relationship
SKIN INDURATION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Any Relationship
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Any Relationship
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — Any Relationship
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — Any Relationship
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Any Relationship
DERMATITIS ACNEFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Any Relationship
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Any Relationship
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Any Relationship
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Any Relationship
DIZZINESS (Nervous system disorders) | 2 | 0 | 1 | 5 — Any Relationship
AGEUSIA (Nervous system disorders) | 1 | 0 | 0 | 0 — Any Relationship
ATAXIA (Nervous system disorders) | 1 | 0 | 0 | 0 — Any Relationship
CONVULSION (Nervous system disorders) | 1 | 0 | 0 | 0 — Any Relationship
HEADACHE (Nervous system disorders) | 1 | 3 | 0 | 4 — Any Relationship
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0 | 0 — Any Relationship
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 1 | 0 | 0 | 0 — Any Relationship
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 1 | 0 | 5 — Any Relationship
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0 — Any Relationship
TREMOR (Nervous system disorders) | 1 | 0 | 0 | 1 — Any Relationship
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0 | 0 — Any Relationship
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 1 | 4 — Any Relationship
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1 | 0 | 0 — Any Relationship
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 1 | 0 — Any Relationship
DIZZINESS POSTURAL (Nervous system disorders) | 0 | 0 | 0 | 1 — Any Relationship
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 1 — Any Relationship
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 0 | 1 — Any Relationship
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 1 — Any Relationship
HAEMATURIA (Renal and urinary disorders) | 2 | 2 | 0 | 3 — Any Relationship
POLLAKIURIA (Renal and urinary disorders) | 2 | 0 | 0 | 1 — Any Relationship
PROTEINURIA (Renal and urinary disorders) | 1 | 0 | 0 | 3 — Any Relationship
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 1 | 1 — Any Relationship
DYSURIA (Renal and urinary disorders) | 0 | 2 | 0 | 2 — Any Relationship
BLADDER PAIN (Renal and urinary disorders) | 0 | 0 | 1 | 1 — Any Relationship
RENAL INJURY (Renal and urinary disorders) | 0 | 0 | 1 | 0 — Any Relationship
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 3 — Any Relationship
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 | 0 | 0 | 1 — Any Relationship
LEUKOCYTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 — Any Relationship
POLYURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 — Any Relationship
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 1 — Any Relationship
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0 | 0 | 1 — Any Relationship
NEUTROPHIL COUNT INCREASED (Investigations) | 1 | 0 | 0 | 0 — Any Relationship
WEIGHT DECREASED (Investigations) | 1 | 4 | 1 | 0 — Any Relationship
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 0 | 1 | 1 — Any Relationship
BLOOD CREATININE INCREASED (Investigations) | 0 | 1 | 1 | 0 — Any Relationship
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 1 | 0 | 0 — Any Relationship
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1 | 1 — Any Relationship
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 1 — Any Relationship
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 0 | 1 — Any Relationship
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 — Any Relationship
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 1 — Any Relationship
URINE OUTPUT DECREASED (Investigations) | 0 | 0 | 0 | 1 — Any Relationship
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 — Any Relationship
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 — Any Relationship
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 4 — Any Relationship
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 — Any Relationship
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 — Any Relationship
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 — Any Relationship
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 — Any Relationship
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 — Any Relationship
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — Any Relationship
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 — Any Relationship
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 — Any Relationship
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 | 0 | 0 | 0 — Any Relationship
CYTOLYTIC HEPATITIS (Hepatobiliary disorders) | 1 | 0 | 1 | 1 — Any Relationship
HEPATOBILIARY DISEASE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 — Any Relationship
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 1 | 0 | 0 | 0 — Any Relationship
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Any Relationship
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Any Relationship
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Any Relationship
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 — Any Relationship
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 — Any Relationship
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 — Any Relationship
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 — Any Relationship
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — Any Relationship
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 — Any Relationship
SNAKE BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 — Any Relationship
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 1 | 1 — Any Relationship
INSOMNIA (Psychiatric disorders) | 1 | 3 | 3 | 2 — Any Relationship
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 1 — Any Relationship
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 0 — Any Relationship
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 1 | 0 — Any Relationship
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 1 | 0 — Any Relationship
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 2 — Any Relationship
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 1 — Any Relationship
SCROTAL DISORDER (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 — Any Relationship
PENIS DISORDER (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 — Any Relationship
HAEMORRHAGE (Vascular disorders) | 1 | 0 | 0 | 0 — Any Relationship
HYPOTENSION (Vascular disorders) | 1 | 0 | 1 | 1 — Any Relationship
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 1 — Any Relationship
EMBOLISM (Vascular disorders) | 0 | 1 | 0 | 0 — Any Relationship
FLUSHING (Vascular disorders) | 0 | 1 | 1 | 0 — Any Relationship
HAEMATOMA (Vascular disorders) | 0 | 0 | 1 | 0 — Any Relationship
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 0 — Any Relationship
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 3 — Any Relationship
HYPOTHYROIDISM (Endocrine disorders) | 0 | 1 | 0 | 0 — Any Relationship
DRY EYE (Eye disorders) | 0 | 1 | 0 | 0 — Any Relationship
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 1 | 1 — Any Relationship
BLEPHAROSPASM (Eye disorders) | 0 | 0 | 0 | 1 — Any Relationship
BLINDNESS UNILATERAL (Eye disorders) | 0 | 0 | 0 | 1 — Any Relationship
CATARACT (Eye disorders) | 0 | 0 | 0 | 1 — Any Relationship
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 1 — Any Relationship
EYE INFLAMMATION (Eye disorders) | 0 | 0 | 0 | 1 — Any Relationship
SINUS OPERATION (Surgical and medical procedures) | 0 | 1 | 1 | 0 — Any Relationship
CENTRAL VENOUS CATHETER REMOVAL (Surgical and medical procedures) | 0 | 0 | 1 | 0 — Any Relationship

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less